CLINICAL TRIAL: NCT04134182
Title: A Phase 2 Pilot Study of the Efficacy and Safety of Nivolumab and Ipilimumab in T1aN0M0 Renal Cell Carcinoma Patients Ineligible for Surgical Treatment.
Brief Title: Nivolumab and Ipilimumab in T1aN0M0 Renal Cell Carcinoma Patients Ineligible for Surgical Treatment.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCRB16102019
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Ipilimumab (Experimental): Patients will receive a combination of ipilimumab, followed by nivolumab for 16 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg intravenously every 2 weeks during 16 weeks
  Other Names: Opdivo
Drug: Ipilimumab — 1 mg/kg intravenously every 3 weeks for four doses
  Other Names: Yervoy

SUMMARY:
The aim of this Phase 2 study is to evaluate the efficacy and safety of nivolumab, an anti-PD-1 antibody, and ipilimumab, an anti-CTLA-4 antibody, in T1aN0M0 clear-cell RCC patients ineligible for surgical treatment.

DETAILED DESCRIPTION:
Surgery remains the standard curative-intent therapy for localized renal cell carcinoma (RCC). Thus, systemic therapy for RCC should still be considered only in patients who have contraindications to surgery.

Results of Phase 3 CheckMate 214 study showed that a combination of nivolumab and ipilimumab has a significant impact on tumor burden in intermediate- and poor-risk metastatic RCC patients with a complete response rate of 11% (Motzer et al. Lancet Oncology 2019). Median time to objective response was 2.8 months. Among all complete responders to nivolumab plus ipilimumab in the intention-to-treat population, 5% achieved a complete response at the first scan, whereas most converted from the partial response at a median of 6.9 months or from the stable disease at a median of 11.3 months.

We hypothesize that this combination could completely eliminate primary tumors in patients with small primary (less than 4 cm) ineligible for surgical treatment. There are no studies evaluating checkpoint inhibitors in this setting in RCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically proven clear-cell RCC
2. CT-confirmed measurable primary tumor less than 4 cm and no evidence of extranodal metastatic disease (T1aN0M0)
3. Inability to perform surgery for any reason (functional single kidney with a central, high-complexity RCC, high risk of nephrectomy and dialysis, patients with complex coagulation disorders, etc.) or preference of patient is to have no surgery for any reason
4. No contradictions to nivolumab and ipilimumab
5. Age 18 or older
6. Written informed consent

Exclusion Criteria:

1. prior treatment for RCC
2. pregnant or nursing
3. history of serious hypertension, cardiac arrhythmia, congestive heart failure, angina pectoris, or another severe cardiovascular disease (i.e., New York Heart Association class III or IV)
4. evidence of metastatic disease
5. local and/or systemic infections requiring antibiotics within 28 days prior to study entry
6. other malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | 16 weeks
  percentage of patients with localized RCC who have no tumor in kidney

SECONDARY OUTCOMES:
Objective response rate | 16 weeks
  percentage of patients with localized RCC who have no tumor in kidney or tumor shrinkage more than 30%
3-year disease-free survival rate | 3 years
  percentage of patients who are disease free at 3 years after treatment start
5-year survival rate | 5 years
  percentage of patients who are alive at 5 years after treatment start
Rate of adverse events | 16 weeks
  percentage of patients who have adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Tsimafeyeu, MD, Study Director — Kidney Cancer Research Bureau
Locations (2):
- Russia (2):
  - N.N. Blokhin Russian Cancer Research Center, Moscow
  - Russian Scientific Center of Roentgenoradiology, Moscow

IPD SHARING:
Plan to Share IPD: No